CLINICAL TRIAL: NCT03889574
Title: Triple Antithrombotic Therapy in Cardiac Patients Requiring Revascularization
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 071.PHA.2018.D
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Disease
Keywords: ICD10 for ACS, STEMI or NSTEMI, Atrial Fibrillation
MeSH Terms: conditions — Heart Diseases; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- combination of aspirin, P2Y12 Inhibitor with a NOAC: As this is a retrospective study with limited patients available for the cohort, all patients meeting inclusion criteria from April 1, 2017 - April 1, 2018 will be included to obtain the largest sample size possible
- combination of aspirin, P2Y12 Inhibitor with warfarin: As this is a retrospective study with limited patients available for the cohort, all patients meeting inclusion criteria from April 1, 2017 - April 1, 2018 will be included to obtain the largest sample size possible

SUMMARY:
Aim(s)/Objective(s)

* To evaluate the safety and efficacy of triple antithrombotic therapy in patients taking DAPT of aspirin and a P2Y12 inhibitor in addition to either a NOAC or warfarin for the prevention of thromboembolic or acute coronary syndrome (ACS) events in patients with non-valvular atrial fibrillation (AF), history of coronary artery disease (CAD)/stent placement or recurrent ACS event.
* To determine the Methodist Health System (MHS) prescribing practices and patterns in cardiac patients with a history of AF who are admitted for CAD or an ACS event requiring PCI.

Hypothesis Primary Hypothesis Cardiac patients with a history of AF and an indication for long-term NOAC who are also prescribed DAPT following an ASC event or revascularization with stenting will demonstrate a significant difference in cardiovascular outcomes and major bleeding events when compared with warfarin-based triple therapy.

DETAILED DESCRIPTION:
STUDY DESIGN

* Multi-center, retrospective cohort chart review study design
* Data will be collected on all triple therapy recipients who were discharged from a Methodist Health System (MHS) facility with prescriptions for a combination of aspirin, P2Y12 Inhibitor and an OAC of either a NOAC or warfarin between April 1, 2017 - April 1, 2018
* Patient list will be generated in EPIC
* All data will be obtained from EPIC
* All data will be collected retrospectively after the patient is discharged from the hospital
* Data collection (planned completion date): May 2019

Study Inclusion Criteria:

* 18 years or older
* AF diagnosis
* ICD10 for ACS, STEMI or NSTEMI
* Discharged with triple therapy agents of aspirin, P2Y12 inhibitor (clopidogrel, prasugrel, or ticagrelor), and OAC (warfarin, edoxaban, dabigatran, rivaroxaban, or apixaban) status post-stent

Study Exclusion Criteria:

* Patients less than 18 years of age
* Prior intracranial bleeding prior to study start date
* GI hemorrhage within 1 month prior to study start date
* Major bleeding event with 1 month prior to study start date
* Hemorrhage disorder
* Stroke within 1 month prior to study start date
* Cardiogenic shock during admission at start date
* Contraindication to use of the study medications
* Peptic ulcer in the prior 6 months prior to study start date
* Thrombocytopenia (platelet concentration lower than 50×109/L)
* Thrombolysis In Myocardial Infarction (TIMI) major bleeding in the prior 12 months of study start date
* Pregnancy
* History of DVT or PE currently on OAC

ELIGIBILITY:
Inclusion Criteria:

* • 18 years or older

  * AF diagnosis
  * ICD10 for ACS, STEMI or NSTEMI
  * Discharged with triple therapy agents of aspirin, P2Y12 inhibitor (clopidogrel, prasugrel, or ticagrelor), and OAC (warfarin, edoxaban, dabigatran, rivaroxaban, or apixaban) status post-stent

Exclusion Criteria:

* • Patients less than 18 years of age

  * Prior intracranial bleeding prior to study start date
  * GI hemorrhage within 1 month prior to study start date
  * Major bleeding event with 1 month prior to study start date
  * Hemorrhage disorder
  * Stroke within 1 month prior to study start date
  * Cardiogenic shock during admission at start date
  * Contraindication to use of the study medications
  * Peptic ulcer in the prior 6 months prior to study start date
  * Thrombocytopenia (platelet concentration lower than 50×109/L)
  * Thrombolysis In Myocardial Infarction (TIMI) major bleeding in the prior 12 months of study start date
  * Pregnancy
  * History of DVT or PE currently on OAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac patients with a history of AF and an indication for long-term NOAC who are also prescribed DAPT following an ASC event or revascularization with stenting
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Comparison between warfarin based triple therapy versus NOAC-based triple therapy in cardiac patients | April 1, 2017 - April 1, 2018
  To compare the incidence of MACE, stroke (ischemic and hemorrhage), MI (STEMI and NSTEMI), stent thrombosis, systemic embolism (VTE), death (all-cause, cardiac and non-cardiac) and CAD-associated hospitalizations/ED visits) in patients who received warfarin-based triple therapy versus NOAC-based triple therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Hansen ML, Sorensen R, Clausen MT, Fog-Petersen ML, Raunso J, Gadsboll N, Gislason GH, Folke F, Andersen SS, Schramm TK, Abildstrom SZ, Poulsen HE, Kober L, Torp-Pedersen C. Risk of bleeding with single, dual, or triple therapy with warfarin, aspirin, and clopidogrel in patients with atrial fibrillation. Arch Intern Med. 2010 Sep 13;170(16):1433-41. doi: 10.1001/archinternmed.2010.271. PMID 20837828